CLINICAL TRIAL: NCT04677218
Title: Comparison of Clinical Results of Adjustable Femoral Loop With Three Different Techniques in Patients Who Underwent Arthroscopic ACL Reconstruction With Hamstring Autograft: A Prospective Randomised Clinical Study
Brief Title: Prospective Clinical Results of 3 Different Femoral Fixation in ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emre Kocazeybek (Other)
Responsible Party: Sponsor-Investigator, Emre Kocazeybek, Resident in the orthopedics and Traumatology department, Istanbul University
Organization: Istanbul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 67990154
Record Dates: First submitted 2020-12-17; First posted 2020-12-21 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: ACL Injury; Anterior Cruciate Ligament Rupture
Keywords: ACL injury; Adjustable femoral loop; Arthroscopic ACL reconstruction; outcomes
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First Group (No Intervention): First group of fixation will be standar procedure ( without knotted and retensioned the hamstring autograft after tibial fixation)
- Second Group (Experimental): In the second group, the hamstring autograft will be retensioned after tibial fixation.
  Interventions: Procedure: Arthroscopic ACL reconstruction with retensioned hamstring autograft
- Third Group (Active Comparator): In the third group, the hamstring autograft will be knotted and retensioned after tibial fixation.
  Interventions: Procedure: Arthroscopic ACL reconstruction with retensioned and knotted hamstring autograft

INTERVENTIONS:
Procedure: Arthroscopic ACL reconstruction with retensioned hamstring autograft — After diagnostic arthroscopy, an oblique, 5-cm oblique skin incision is made below the joint line over the proximal edge of the pes anserine.Then fascia will be incised the fascia in an L-shaped fashion. After the releasing the distal end of tendons ,tendons will be harvested in their direction via tendon strippers.During the graft preparation phase firstly femoral tunel will be drilled from AM portal with knee flexed to 120 degrees. The drill will be aligned parallel to the tibial plateau and exit through LFC.Then tibial guide wire will be sent from graft incision to the tibial tunel and drilled for desired direction.Once the adjustable loop button is deployed to the graft, it will be pulled through the tunnels and the button is slipped on lateral femoral cortex. Then tibial fixation will be provided with one bioabsorbable screw and staple.After tibial fixation, the femoral loop will be retensioned in group 2 patients.
  Arms: Second Group
Procedure: Arthroscopic ACL reconstruction with retensioned and knotted hamstring autograft — After the same preparation procedure as in retensioned autograft group, after tibial fixation of graft, femoral loop will be retensioned and knotted in 3. group .
  Arms: Third Group

SUMMARY:
Anterior cruciate ligament (ACL) tears are one of the most common injuries of the knee. In today's world, due to developing sports industry , the increase in sports traumas of both genders and ages ACL injuries and treatments are given major priority.

The success of anterior cruciate ligament (ACL) reconstruction depends on many factors, including the mechanical properties of the graft, positioning of the proper femoral and tibial tunnel, fixation methods and the postoperative rehabilitation.

The tendon grafts can be fixed on the femoral side using several fixation devices, including cortical suspension devices, cross pins, and interference screws. Femoral fixation via Cortical button in a suture loop provides the highest primary stability, and therefore, has become increasingly popular among orthopaedic surgeons. Adjustable and fixed Femoral cortical loops are commonly used for femoral fixation. In this sudy we aimed to compare clinical and functional outcomes of three different techniques of suspensory femoral fixation in ACL reconstruction.

DETAILED DESCRIPTION:
This study has been planned as a prospective randomized clinical trial. We used a completely computer-generated list in order to randomize all participants to receive one of two treatments (www.random.org/sequences/).

Anterior Cruciate Ligament tear diagnosis will be made by physical examination and magnetic resonance imaging. Participants who agree to be enrolled to study will be examined one day prior to surgery. Patients are randomly divided into 3 groups, after tibial fixation of the hamstring autograft, 3 different techniques will be used in the femoral fixation phase.

The first group will be without knotting and retensioning the graft. In the second group, The graft will be retensioned after tibial fixation. In the third group femoral loop will be retensioned and knotted after tibial fixation.

All the surgeries will be performed by the same senior surgeon experienced in sports medicine surgery under regional anesthesia with patient in supine position.

All participants will receive a standard postoperative rehabilitation program starting immediately after surgery with closed chain exercises and quadriceps strengthening and walking. The operated lower extremity won't be placed in a brace and patient allowed for full weight walking with a pair of crutches.

Postoperative evaluations will be performed regularly at 12 months postoperatively . To assess knee stability, KT-1000 measurement will be applied to both extremities in each group and clinical scores ( lysholm knee score, IKDC ) will be measured.

Furthermore, to evaluate flexor and extensor muscle group around knee, isokinetic tests will be applied to patients in sitting position to analyse peak torque and total work done values.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ACL Rupture between the ages of 18-55
* Patients with isolated + primary ACL rupture only
* Patients with ACL rupture ± meniscal tear

Exclusion Criteria:

* Patients with Posterior cruciate ligament rupture
* Multiligamentous knee injuries
* Patients with Medial or Lateral Collateral injuries
* Patients with previous revision surgeries

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Kt-1000 Stability | 12.months postoperatively
  The KT1000 arthrometer is designed to measure the anterior translation of the tibia while maintaing the femur in position. The results obtained provide an objective diagnostic of the state of the ACL. The healthy leg will be tested first followed by the injured leg. The side-to-side differences will be then evaluated at each force, which allows the diagnosis of the knee laxity.
Isokinetic Knee tests | 12.months postoperatively
  Flexor and Extansor muscle group of the knee

SECONDARY OUTCOMES:
IKDC scores | 12.months postoperatively
  Determining of knee symptoms Function, and activity of daily living
Tegner-Lysolm score | 12.months postoperatively
  This is a clinical functional assessment test used for Ligamentous knee disorders. Including 8 parameters .
Postoperative Range of motion | 6.months and 12.months postoperatively
  Knee flexion, Extension will be masured by goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan Polat, M.D, Principal Investigator — Istanbul University Istanbul Medical Faculty
Locations (1):
- Istanbul University Istanbul Medical Faculty Department of Orthopedics and Traumatology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi NH, Yang BS, Victoroff BN. Clinical and Radiological Outcomes After Hamstring Anterior Cruciate Ligament Reconstructions: Comparison Between Fixed-Loop and Adjustable-Loop Cortical Suspension Devices. Am J Sports Med. 2017 Mar;45(4):826-831. doi: 10.1177/0363546516674183. Epub 2016 Nov 25. PMID 27881383
- [Background] Ahn HW, Seon JK, Song EK, Park CJ, Lim HA. Comparison of Clinical and Radiologic Outcomes and Second-Look Arthroscopic Findings After Anterior Cruciate Ligament Reconstruction Using Fixed and Adjustable Loop Cortical Suspension Devices. Arthroscopy. 2019 Jun;35(6):1736-1742. doi: 10.1016/j.arthro.2019.01.051. Epub 2019 May 6. PMID 31072714
- [Background] Onggo JR, Nambiar M, Pai V. Fixed- Versus Adjustable-Loop Devices for Femoral Fixation in Anterior Cruciate Ligament Reconstruction: A Systematic Review. Arthroscopy. 2019 Aug;35(8):2484-2498. doi: 10.1016/j.arthro.2019.02.029. Epub 2019 May 27. PMID 31147109
- [Background] Boyle MJ, Vovos TJ, Walker CG, Stabile KJ, Roth JM, Garrett WE Jr. Does adjustable-loop femoral cortical suspension loosen after anterior cruciate ligament reconstruction? A retrospective comparative study. Knee. 2015 Sep;22(4):304-8. doi: 10.1016/j.knee.2015.04.016. Epub 2015 May 19. PMID 25999126
- [Background] Tegner Y, Lysholm J. Rating systems in the evaluation of knee ligament injuries. Clin Orthop Relat Res. 1985 Sep;(198):43-9. PMID 4028566
- [Result] Choi NH, Victoroff BN. Author Reply to "Regarding 'Radiologic and Clinical Outcomes After Hamstring Anterior Cruciate Ligament Reconstruction Using an Adjustable-Loop Cortical Suspension Device With Retensioning and Knot Tying'". Arthroscopy. 2020 Apr;36(4):931-933. doi: 10.1016/j.arthro.2020.01.028. No abstract available. PMID 32247421
- See also: Web site used for randomization of participants — https://www.random.org/sequences/